CLINICAL TRIAL: NCT00763048
Title: Collection of Gingival Crevicular Fluid From Periodontitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRO-2007-GIN-05-GB
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases | interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A -Control (Placebo Comparator): Fluoride toothpaste (Colgate Great Regular Flavor) is the control for this study. All study toothpastes contain fluoride. The study is evaluating the additional ingredients in the other toothpastes.
  Interventions: Drug: Fluoride
- B (Active Comparator): fluoride/triclosan/copolymer toothpaste (Colgate Total Toothpaste)
  Interventions: Drug: Fluoride, triclosan

INTERVENTIONS:
Drug: Fluoride — Brush twice daily for 6 weeks
  Other Names: Coglate Great Regular Flavor toothpaste
  Arms: A -Control
Drug: Fluoride, triclosan — Brush twice daily
  Other Names: Colgate Total toothpaste
  Arms: B

SUMMARY:
To collect GCF (gingival crevicular fluid) samples from diseased patients suffering only from gingivitis and/or periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 to 65 years inclusive
* Have a minimum of 20 natural uncrowned teeth (excluding 3rd molars) present
* Give written informed consent
* Be in good general health
* No known history of allergy to personal care/consumer products or their
* ingredients, relevant to any ingredients in the test products as determined by the
* dental/medical professional monitoring the study

Exclusion Criteria:

* Medical condition which requires pre-medication prior to dental visits/procedures
* Advanced periodontal disease
* 5 or more decayed, untreated dental sites
* Diseases of the soft or hard oral tissues
* Orthodontic appliances
* Abnormal salivary function
* Use of prescription drugs.
* Use of antibiotics one (1) month prior to or during this study
* Use of any over the counter medications other than analgesics
* Erratic use of vitamin supplements
* Pregnant or breastfeeding.
* Participation in another clinical study in the month preceding this study
* Allergic to common dentifrice ingredients
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 26 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Teles, DMD, Principal Investigator
Locations (1):
- Forsyth Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Pre-assignment Details: Subjects were screened to meet medical and oral health criteria and then began a 1 week washout period with fluoride toothpaste.
Groups:
- A - Control Comparator: Participants brushed their teeth with the fluoride only control toothpaste two times a day for six weeks.
- B - Active Comparator: Participants rinsed their teeth with the Active Comparator toothpaste (fluoride/triclosan/copolymer) two times a day for six weeks.
Period: Overall Study
Arm/Group | A - Control Comparator | B - Active Comparator
Started | 21 | 18
Completed | 21 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Control Comparator | B - Active Comparator | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (12.7) | 49.8 (12.8) | 48.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Metabolite Associated With Inflammation (Cadaverine)
Description: One of 10 inflammation biomarkers found in gingival crevicular fluid (GCF) that are associated with inflammation that could lead to gingivitis. The number is a quantitative, normalized ion count from a mass spectral instrument. The lower the number the less inflammation may be present. Data is after 6 weeks use of the study treatment.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.119186 (0.834969) | 0.92077 (0.78476)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Primary Outcome: Metabolite Associated With Inflammation (Choline)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.2264 (0.79066) | 1.169513 (0.79071)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

3. Primary Outcome: Metabolite Associated With Inflammation (Hypoxanthine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 0.76984 (0.58459) | 0.701628 (0.63887)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

4. Primary Outcome: Metabolite Associated With Inflammation (Inosine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.11183 (1.05685) | 0.84462 (0.99409)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

5. Primary Outcome: Metabolite Associated With Inflammation (Isoleucine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.20033 (0.61108) | 1.048449 (0.70947)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

6. Primary Outcome: Metabolite Associated With Inflammation (Leucine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.10064 (0.5424) | 1.018989 (0.64132)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

7. Primary Outcome: Metabolite Associated With Inflammation (Lysine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.063873 (0.785917) | 1.09704 (1.149168)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

8. Primary Outcome: Metabolite Associated With Inflammation (Phenylalanine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.16994 (0.56433) | 1.057373 (0.625110)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

9. Primary Outcome: Metabolite Associated With Inflammation (Putrescine)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.050398 (0.69913) | 0.74134 (0.86837)
Statistical Analysis 1: Comparison: A - Control Comparator vs B - Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

10. Primary Outcome: Metabolite Associated With Inflammation (Xanthine)
Description: One of 10 inflammation biomarkers found in gingival crevicular fluid (GCF) that are associated with inflammation that could lead to gingivitis. The number is a quantitative, normalized ion count from a mass spectral instrument. The lower the number the less inflammation may be present.Data is after 6 weeks use of the study treatment.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ion count
Arm/Group | A - Control Comparator | B - Active Comparator
Number analyzed (Participants) | 21 | 18
ion count | 1.05189 (0.615226) | 1.011732 (0.96834)

ADVERSE EVENTS:
Time Frame: 7 weeks (1 week washout period + 6 week study treatment period)
Arm/Group | A - Control Comparator | B - Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less